CLINICAL TRIAL: NCT02171793
Title: A Randomised, Single-blind, Placebo-controlled (Within Dose Groups) Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Peroral Doses (15, 30, 40 μg Free Cation) BI 1744 CL in Healthy Male Volunteers
Brief Title: Single Rising Peroral Doses of BI 1744 CL in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1222.19
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — olodaterol

ARMS (2):
- BI 1744 CL (Experimental)
  Interventions: Drug: BI 1744 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1744 CL
  Arms: BI 1744 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate safety, tolerability, and pharmacokinetics of single rising peroral doses of BI 1744 CL.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥21 and ≤45 years
* BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
* Evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomisation
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug within 30 days prior to randomisation
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days as judged by the investigator
* Alcohol abuse (regularly more than 40 g alcohol per day)
* Drug abuse
* Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
* Excessive physical activities within 1 week prior to randomisation or during the trial
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of the study centre

The following exclusion criteria are specific for this study due to the known class side effect profile of β2 mimetic drugs:

* Asthma or history of pulmonary hyperreactivity
* Hyperthyrosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia
* Paroxysmal tachycardia (>100 beats per minute)

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline, day 17
Number of patients with clinically significant changes in vital signs (blood pressure (BP), pulse rate (PR), respiration rate (RR), oral body temperature) | Baseline, up to day 17
Number of patients with clinically relevant abnormal findings in 12-lead electrocardiogram (ECG) | Baseline, up to day 17
Number of patients with clinically significant changes in clinical laboratory tests | Baseline, up to day 17
Number of patients with Adverse events (AEs) | 5 weeks
Assessment of tolerability by investigator on a 4-point scale | Day 17

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
λz (terminal rate constant in plasma) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
MRTpo (mean residence time of the analyte in the body after peroral administration) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
CL/F (apparent clearance of the analyte in plasma after peroral administration, will not be calculated for metabolites) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following a peroral dose, will not be calculated for metabolites) | pre-dose and 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | pre-dose and 0-4, 4-8, 8-12, 12-24, 24-48 h after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | pre-dose and 0-4, 4-8, 8-12, 12-24, 24-48 h after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | pre-dose and 0-4, 4-8, 8-12, 12-24, 24-48 h after drug administration